CLINICAL TRIAL: NCT06577623
Title: In-Person Mindfulness-based Intervention for Adolescents with Autism Spectrum Disorder and Their Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southwest Autism Research & Resource Center (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00016672b
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Open label feasibility and acceptability trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MINDful TIME group (Experimental): 8-week mindfulness-based intervention for adolescents with ASD and their caregivers. Weekly meetings will be held in-person and will last approximately 2-hours. Adolescents and their caregivers will be asked to engage in home practice outside of group meetings
  Interventions: Behavioral: MINDful TIME

INTERVENTIONS:
Behavioral: MINDful TIME — Group-based psychoeducational mindfulness-based intervention.

SUMMARY:
Adolescents with ASD often have co-occurring mental health symptoms like stress, anxiety, and depression. The investigators are conducting this research study to develop interventions for adolescents with ASD that will improve co-occurring mental health symptoms.

DETAILED DESCRIPTION:
Adolescents with ASD and their parents will complete a 3-hour in-person screening visit to determine eligibility for the study.

Adolescents with ASD and their caregivers will participate in an 8-week mindfulness-based group intervention that meets once weekly at SARRC in Phoenix, Arizona. Each meeting will last approximately 2-hours. Teens and parents/caregivers will have separate meetings with separate group leaders but will reunite for approximately 15-minutes as a larger group to review home practice for the upcoming week. Teens and parents will each be given a free 1-year subscription to Ten Percent Happier, a commercially available mobile app focused on mindfulness meditations. Each week teens will be assigned home practice, which means we will ask participants to practice mindfulness meditation every day. The investigators will recommend specific meditations and activities to complete, but participants will have access to all mindfulness meditations on the Ten Percent Happier app.

Teens and caregivers will be asked to complete questionnaires assessing things like mood, anxiety, quality of life, mindfulness in day-to-day life, and their perception of the intervention. These questionnaires will be done immediately before the intervention, immediately after completing the intervention, and at 2-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents must be ages 13 to 18 years
* Formal clinical or educational ASD diagnosis confirmed by the study team (i.e., review of the formal diagnostic or educational report)
* Must be able to attend at least 7 of the 8 in-person group meetings
* English speaking: Adolescents and their parent/caregivers must be English-speaking because the screening and behavioral measures are in English, as well as the intervention content

Exclusion Criteria:

* Non-verbal participants will be excluded to ensure test compliance and increase sample homogeneity.
* Participants with IQ scores <70 will be excluded because the intervention was developed for individuals without intellectual disabilities.
* Participants with a physical disability or co-occurring condition that may prevent participation in the weekly group meetings (e.g., selective mutism; aggressive behavior; inability to participate in a 90-minute video conference meeting each week)
* Participants who report active suicidal ideation

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in Children's Depression Inventory (CDI) Scores | Post-intervention (8 weeks); 2-month follow-up
  Parent-report measure of adolescent depressive symptoms. Scores range from 30 to 90 with higher scores indicating higher levels of depression symptoms.
Mean Change from Baseline in Multidimensional Anxiety Scale for Children (MASC) Scores | Post-intervention (8 weeks); 2-month follow-up
  Parent-report measure of adolescent anxiety symptoms. Scores range from 30 to 90 with higher scores indicating higher levels of anxiety symptoms.
Mean Change from Baseline in Child and Adolescent Mindfulness Measure (CAMM) Scores | Post-intervention (8 weeks); 2-month follow-up
  Adolescent-report measure of mindfulness. Scores range from 0 to 40 with higher scores indicating higher levels of mindfulness.

SECONDARY OUTCOMES:
Mean Change from Baseline in Beck Youth Inventories (BYI) Scores | Post-intervention (8 weeks); 2-month follow-up
  Adolescent-report measure of depression. Scores range from 0 to 90, with higher scores indicating higher levels of depression.
Mean Change from Baseline in World Health Organization-Five Wellbeing Index (WHO-5) Scores | Post-intervention (8 weeks); 2-month follow-up
  Adolescent-report measure on current well-being. Scores range from 0 to 100, with higher scores indicating better quality of life.
Mean Change from Baseline in Adaptive Behavior Assessment System (ABAS-3) Scores | Post-intervention (8 weeks); 2-month follow-up
  Parent-report measure of adolescent adaptive skills across the lifespan. Scores range from 40 to 120, with higher scores indicating better adaptive skills.
Mean Change from Baseline in Behavior Rating Inventory of Executive Function (BRIEF) Scores | Post-intervention (8 weeks); 2-month follow-up
  Parent-report measure of adolescent executive function and self-regulation. Scores range from 30 to 90, with higher scores indicating higher levels of executive dysfunction.
Mean Change from Baseline in Five Facets Mindfulness Questionnaire (FFMQ) Scores | Post-intervention (8 weeks); 2-month follow-up
  Adolescent-report measure of mindfulness on observation, description, aware actions, non-judgmental inner experience, and non-reactivity. Factor scores range from 1 to 5, with higher scores indicating higher levels of mindfulness.
Mean Change from Baseline in Stress Index for Parents of Adolescents (SIPA) Scores | Post-intervention (8 weeks); 2-month follow-up
  Parent-report measure of the relationship of parenting stress to adolescent characteristics, parent characteristics, the quality of the adolescent-parent interactions, and stressful life circumstances. Percentile scores range from 0 to 99, with higher scores indicating higher levels of parenting stress.
Mean Change from Baseline in Social Responsiveness Scale (SRS-2) Scores | Post-intervention (8 weeks); 2-month follow-up
  Parent-report measure of adolescent presence and severity of social impairment within autism spectrum. T-scores range from 30 to > 90 with higher scores indicating greater social impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Matthews, Ph.D., Principal Investigator — Southwest Autism Research & Resource Center
Locations (1):
- Southwest Autism Research and Resource Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided